CLINICAL TRIAL: NCT06020313
Title: Evaluation of the Metabolic Profile and Autonomic and Cardiovascular Recovery in Response to the Acute Use of Resveratrol in Individuals With Overweight and Obesity
Brief Title: Autonomic and Cardiovascular Recovery After the Acute Use of Resveratrol in Overweight and Obesity Individuals
Acronym: Resveratrol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taisy Cinthia Ferro Cavalcante (Other)
Responsible Party: Sponsor-Investigator, Taisy Cinthia Ferro Cavalcante, doctor, University of Pernambuco
Organization: University of Pernambuco (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 5.051.852
Record Dates: First submitted 2023-06-26; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Polyphenols; Cardiovascular Diseases; Autonomic Nervous System
Keywords: Resveratrol; Cardiovascular Diseases; Autonomic Nervous System
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This research is a randomized, double-blind, crossover, placebo-controlled clinical trial. Volunteers of both sexes aged between 20 and 59 years, with overweight or obesity grade I. Therefore, on the first day of collection, volunteers will be allocated to one of the following treatment protocols: Protocol I) Placebo or Protocol II) Experimental (Resveratrol, 500 mg). After ingestion, the heart rate receiver Polar RS800CX (Polar Electro, Finland) will be positioned on the chest of the volunteers. The blood pressure of the participants will be measured before (Rest) and after the submaximal strength exercise, during the first recovery time (REC1- 00-05 minutes) in 5 intervals, using an aneroid sphygmomanometer and stethoscope. Participants will be previously informed about blood collection for the evaluation of the biochemical profile of the following serum analytes: glucose, triglycerides, total cholesterol and fractions, albumin, total proteins and uric acid.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers who will do the experiment will be blind. They will not know who is the experimental group and the control group. The distribution of groups will be carried out by a partner researcher who is part of our research group, but is not directly involved in the current research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Resveratrol (Experimental): Resveratrol capsules (100mg) will be used from 7am to 7pm, de 3 em 3h. That is, at 7 am, 10 am, 1 pm, 4 pm and 7 pm for 7 days.
  Interventions: Dietary Supplement: Resveratrol Experimental
- Placebo (Placebo Comparator): After 48h washout, placebo capsules (100mg) will be used from 7am to 7pm, de 3 em 3h. That is, at 7 am, 10 am, 1 pm, 4 pm and 7 pm for 7 days.
  Interventions: Dietary Supplement: Resveratrol Experimental

INTERVENTIONS:
Dietary Supplement: Resveratrol Experimental — The amount of 500mg per day will be offered for seven days distributed in doses of 100mg per schedule (7am, 10am, 1pm, 4pm and 7pm).

SUMMARY:
The aim of this study is to understand the importance of resveratrol supplementation as a possible adjuvant in improving the metabolic profile and cardiovascular autonomic recovery of individuals with overweight and grade I obesity, reducing the incidence of diseases associated with obesity and the costs in primary, secondary and tertiary care.

DETAILED DESCRIPTION:
Food is a strong ally in improving the metabolic state in overweight, obesity and prevention of associated diseases, working on weight loss and ingestion of anti-inflammatory, anti-oxidant and cardioprotective substances, among these substances, we highlight the polyphenols. Resveratrol or 3,5,4-trihydroxystilbene is a polyphenol studied since 1976, a phytoalexin synthesized in the skin of the grape, which is increased when exposed to stresses such as ultraviolet radiation, enhancing the antioxidant and cardioprotective characteristics.This study aims to evaluate the cardiovascular autonomic recovery and the metabolic profile with the acute effect of resveratrol extract after submaximal aerobic exercises in individuals with overweight and grade I obesity.Heart rate variation (HRV) is considered the most trivial method for analyzing the behavior of autonomic efferents (parasympathetic and sympathetic) on the heart. HRV recovery after exercise has been widely used as a method of analyzing ANS adaptation (vagal recovery) under various conditions.Healthy, physically active individuals with good health characteristics have a rapid recovery of HRV after exercise, indicating good adaptability and a lower risk for cardiovascular diseases. Meanwhile, changes HRV patterns provide a sensitive and early indicator of health impairments. The monitoring of these data is necessary, as they act as markers of emerging risk for the development of complications associated with CNCDs and risks of future injuries. In this context, the present project will make it possible to verify the effect of the acute use of resveratrol on the metabolic profile and on the autonomic and cardiovascular recovery of individuals with overweight and obesity grade I.

ELIGIBILITY:
Inclusion Criteria:

- Individuals with overweight and obesity grade I

Exclusion Criteria:

* Cardiorespiratory disorders
* Neurological disorders
* skeletal muscle injury
* Known impairments that prevent the subject from performing the procedures.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Autonomic and cardiovascular recovery | Five months of collecting and analyzing data.
  Analysis of linear and non-linear indices of heart rate variability
biochemical parameters | Two weeks
  complete blood count, blood glucose, triglycerides, total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Taisy Ferro Cavalcante, Dr, Principal Investigator — University of Pernambuco
Locations (1):
- Taisy Cinthia Ferro Cavalcante, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
This project was approved by the Research Ethics Committee of the University of Pernambuco/CISAM (CEP/UPE-CISAM), opinion number: 5.051.852.
  The results will be published in scientific articles and the final report will be forwarded to the ethics committee.
  Volunteers will be duly informed about the procedures and objectives of this study.
  Before participating, they will sign the Free and Informed Consent Form, being able to withdraw from the study at any time.

REFERENCES:
- [Background] Gonzaga LA, Vanderlei LCM, Gomes RL, Valenti VE. Caffeine affects autonomic control of heart rate and blood pressure recovery after aerobic exercise in young adults: a crossover study. Sci Rep. 2017 Oct 26;7(1):14091. doi: 10.1038/s41598-017-14540-4. PMID 29075019
- [Background] Pecanha T, Bartels R, Brito LC, Paula-Ribeiro M, Oliveira RS, Goldberger JJ. Methods of assessment of the post-exercise cardiac autonomic recovery: A methodological review. Int J Cardiol. 2017 Jan 15;227:795-802. doi: 10.1016/j.ijcard.2016.10.057. Epub 2016 Oct 23. PMID 27836300
- [Background] Tabrizi R , Tamtaji OR , Lankarani KB , Mirhosseini N , Akbari M , Dadgostar E , Peymani P , Asemi Z . The effects of resveratrol supplementation on biomarkers of inflammation and oxidative stress among patients with metabolic syndrome and related disorders: a systematic review and meta-analysis of randomized controlled trials. Food Funct. 2018 Dec 13;9(12):6116-6128. doi: 10.1039/c8fo01259h. PMID 30426122
- [Background] Tome-Carneiro J, Gonzalvez M, Larrosa M, Garcia-Almagro FJ, Aviles-Plaza F, Parra S, Yanez-Gascon MJ, Ruiz-Ros JA, Garcia-Conesa MT, Tomas-Barberan FA, Espin JC. Consumption of a grape extract supplement containing resveratrol decreases oxidized LDL and ApoB in patients undergoing primary prevention of cardiovascular disease: a triple-blind, 6-month follow-up, placebo-controlled, randomized trial. Mol Nutr Food Res. 2012 May;56(5):810-21. doi: 10.1002/mnfr.201100673. PMID 22648627
- [Background] Singh AP, Singh R, Verma SS, Rai V, Kaschula CH, Maiti P, Gupta SC. Health benefits of resveratrol: Evidence from clinical studies. Med Res Rev. 2019 Sep;39(5):1851-1891. doi: 10.1002/med.21565. Epub 2019 Feb 11. PMID 30741437
- [Background] Chekalina NI. Resveratrol has a positive effect on parameters of central hemodynamics and myocardial ischemia in patients with stable coronary heart disease. Wiad Lek. 2017;70(2 pt 2):286-291. PMID 29059644
- [Result] Bastianetto S, Menard C, Quirion R. Neuroprotective action of resveratrol. Biochim Biophys Acta. 2015 Jun;1852(6):1195-201. doi: 10.1016/j.bbadis.2014.09.011. Epub 2014 Oct 2. PMID 25281824
- [Result] Brasnyo P, Molnar GA, Mohas M, Marko L, Laczy B, Cseh J, Mikolas E, Szijarto IA, Merei A, Halmai R, Meszaros LG, Sumegi B, Wittmann I. Resveratrol improves insulin sensitivity, reduces oxidative stress and activates the Akt pathway in type 2 diabetic patients. Br J Nutr. 2011 Aug;106(3):383-9. doi: 10.1017/S0007114511000316. Epub 2011 Mar 9. PMID 21385509